CLINICAL TRIAL: NCT05727891
Title: A Phase 2 Evaluation of Tonabersat for Diabetic Macular Edema (Protocol AN)
Brief Title: Evaluation of Tonabersat for DME
Acronym: AN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRCR Protocol AN; UG1EY014231 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — tonabersat

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Tonabersat (80 mg) (Active Comparator)
  Interventions: Drug: Tonabersat

INTERVENTIONS:
Drug: Tonabersat — Two pills of Study Drug (80 mg tonabersat) is taken orally once daily. It is recommended the Study Drug be taken at bedtime. The first dose (two pills) will be taken at bedtime on the day the participant is randomized.
  Arms: Tonabersat (80 mg)
Other: Placebo — Two pills of Study Drug (placebo) is taken orally once daily. It is recommended the Study Drug be taken at bedtime. The first dose (two pills) will be taken at bedtime on the day the participant is randomized.
  Arms: Placebo

SUMMARY:
This randomized clinical trial will evaluate the effect of tonabersat compared with placebo on central subfield thickness (CST) in eyes with center-involved diabetic macular edema (CI-DME) and good visual acuity.

DETAILED DESCRIPTION:
The primary objective is to assess the effects of tonabersat, an orally administered Connexin43 hemichannel inhibitor, on central subfield thickness (mean change) compared with placebo in eyes with CI-DME and good visual acuity at 6 months.

Exploratory objectives will evaluate biomarkers of kidney function for potential benefit. Furthermore, this phase 2 study is being conducted to determine whether the conduct of a phase 3 trial has merit and provide information on outcome measures needed to design a phase 3 trial.

ELIGIBILITY:
Key Inclusion Criteria

1. Adults with type 1 or 2 diabetes mellitus
2. At least one eye with:

   * Best corrected E-ETDRS visual acuity letter score ≥ 74 (i.e., 20/32 or better)
   * Ophthalmoscopic evidence of center-involved DME in study eye confirmed by central subfield thickness on spectral domain OCT
   * Zeiss Cirrus: ≥ 290 µm in females, ≥ 305 µm in males
   * Heidelberg Spectralis: ≥ 305 µm in females, ≥ 320 µm in males

     * Recruitment will be monitored with a goal to have equal proportions in the following categories above the CI-DME thresholds: <75 μm, 75 μm to <175 μm, ≥175 μm
3. Media clarity, pupillary dilation, and study participant cooperation sufficient for adequate OCT

Key Exclusion Criteria

* Macular edema is considered to be due to a cause other than DME
* Major ocular surgery within prior 4 months, or anticipated after randomization
* History of focal/grid laser or other ocular surgical, intravitreal, or peribulbar treatment for DR or DME within prior 1 year, and no more than 4 anti-VEGF injections within prior 3 years
* Anticipated need to treat DME or DR during the first 6 months, or anticipated need for cataract surgery during study period
* Any history of vitrectomy
* Systemic anti-VEGF or pro-VEGF treatment within 12 months prior to randomization
* History of chronic renal failure requiring dialysis or kidney transplant
* History of moderate to severe hepatic impairment, including known liver function test (LFT) values > 3x's the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in central subfield thickness | 6 months

SECONDARY OUTCOMES:
Mean change in retinal volume from baseline | 6 months
Percentage of eyes central subfield thickness below optical coherence machine- and sex-specific threshold for DME and at least a 10% decrease from baseline | 6 months
  Composite outcome, gender-specific spectral domain optical coherence tomography equivalent of 250 µm on Zeiss Stratus optical coherence tomography
Mean change in visual acuity from baseline | 6 months
Percentage of eyes receiving other treatment for DME prior to the 6 month visit | 6 months

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Retina Associates of Southern California, Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Southern California Desert Retina Consultants, Inc., Palm Desert, California
  - Macula Retina Vitreous Institute, Torrance, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Illinois Retina Associates, Oak Park, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Joseph E. Humble and Raymond Haik PTRS DBA Eye Assoc of Northeast Louisiana, West Monroe, Louisiana
  - Elman Retina Group, Baltimore, Maryland
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Retina Research Institute, LLC, St Louis, Missouri
  - Retina-Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - Verum Research LLC, Eugene, Oregon
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pittsburg Clinical Trial Consortium, Sewickley, Pennsylvania
  - Hilton Head Retina Institute, Hilton Head Island, South Carolina
  - Retina Consultants of Texas, PA, Bellaire, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Retinal Consultants of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No